CLINICAL TRIAL: NCT04576884
Title: Age-Related Changes and Cycloplegia-Induced Differences of the Human Crystalline Lens, Schlemm' s Canal and Trabecular Meshwork：an in Vivo Swept-Source Optical Coherence Tomography Study
Brief Title: Age-Related Changes and Cycloplegia-Induced Differences in the Human Crystalline Lens
Status: Completed | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: SSOCT-ocular parameters change
Record Dates: First submitted 2020-09-21; First posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Cataract
Keywords: radius of curvature; lens thickness; equatorial diameter; lens vault; cycloplegia; swept-source optical coherence tomography; schlemm' s canal; trabecular meshwork
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: participants of less than 18 years old
- Group 2: participants aged from 18 years to 40 year
- Group 3: participants aged from 41 years to 60 years
- Group 4: participants over 60 years old

SUMMARY:
The ocular biometric parameters of the human crystalline lens including anterior chamber depth (ACD), lens thickness (LT), radii of curvature of anterior and posterior lens (ALR and PLR), lens equatorial diameter (LED), and lens vault (LV), automatically quantified by the CASIA2 (SS-OCT; Tomey, Nagoya, Japan). Images of iridocorneal angle were obtained using CASIA2 and the Schlemm' s canal (SC) and trabecular meshwork (TM) were quantified manually. Both cycloplegia and non-cycloplegia images were obtained.

DETAILED DESCRIPTION:
Healthy individuals aged between 6 and 90 years, without history of ocular disease (except age-related cataract and/or myopia), were consecutively included from April to May 2019. All participants underwent visual acuity, dry and wet refraction, anterior and posterior segment examination, intraocular pressure (IOP), and axial length (AL) using IOL-Master 700 (Carl Zeiss Meditec AG). Investigators recruited children under 18 years old at a refraction outpatient clinic, who were prescribed cyclopentolate hydrochloride eyedrops (S.A. Alcon-Couvreur N.V., Belguim) for cycloplegic refraction. For adults, they were prescribed compound tropicamide eyedrops (Mydrin-P, Santen Pharmaceutical Co., Ltd, Osaka, Japan), consisting of 0.5% tropicamide mixed with 0.5% phenylephrine hydrochloride, for pupillary dilation in order to perform fundus examination at an outpatient clinic. Exclusion criteria were as follow:ocular diseases other than cataracts; history of eye surgeries or injuries; shallow anterior chamber with a risk of angle closure. The data from right eye was selected for analysis.

ELIGIBILITY:
Inclusion Criteria:

Healthy individuals aged between 6 and 90 years, without history of ocular disease (except age-related cataract and/or myopia) Must be able to cooperate examination

Exclusion Criteria:

ocular diseases other than cataracts history of eye surgeries or injuries shallow anterior chamber with a risk of angle closure

Ages: 6 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy individuals aged between 6 and 90 years, without history of ocular disease (except age-related cataract and/or myopia) at Eye hospital of Wenzhou Medical University
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Paired Comparison Before and After Cycloplegia | 2020.2.3
  The cycloplegia-induced differences of parameters was defined as: the post-cycloplegic value minus the pre-cycloplegic value.
Evaluated the effect of age on the TM/SC morphologies | 2020.2.3
  The age-related variations of TM/SC parameters from four age groups were compared.

SECONDARY OUTCOMES:
Evaluated the effect of age on the ocular biometric data | 2020.2.3
  The age-related variations of ocular biometric data such as axial length (AL), lens thickness (LT), and anterior chamber depth (ACD) from four age groups were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Yune Zhao, Study Director — Ophthalmology and Optometry Hospital
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Li Z, Meng Z, Qu W, Li X, Chang P, Wang D, Zhao Y. The Relationship Between Age and the Morphology of the Crystalline Lens, Ciliary Muscle, Trabecular Meshwork, and Schlemm's Canal: An in vivo Swept-Source Optical Coherence Tomography Study. Front Physiol. 2021 Nov 19;12:763736. doi: 10.3389/fphys.2021.763736. eCollection 2021. PMID 34867468